CLINICAL TRIAL: NCT05652504
Title: Phase 1 Safety Evaluation of PfSPZ Vaccine in Pregnant Women in Mali (MalVIP1)
Brief Title: Safety Evaluation of PfSPZ Vaccine in Pregnant Women in Mali (MalVIP1)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The study remains on hold due to a funding issue after it's been lifted by the FDA.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10001012; 001012-I
Record Dates: First submitted 2022-12-14; First posted 2022-12-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-16

CONDITIONS: Malaria
Keywords: Immunogenicity; Protective; Efficacy; Tolerability; Randomized
MeSH Terms: conditions — Malaria | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): (n = 30) pregnant women will receive three doses of PfSPZ Vaccine (9x10^5 PfSPZ) via direct venous inoculation (DVI) at 1, 8, 29 days
  Interventions: Biological: PfSPZ Vaccine; Other: PfSPZ Diluent
- Arm 2 (Placebo Comparator): (n = 30) pregnant women will receive normal saline via DVI at 1, 8, 29 days
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — PfSPZ Vaccine contains aseptic, purified, vialed, cryopreserved, radiation attenuated NF54 Pf sporozoites (PfSPZ) produced by Sanaria Inc. PfSPZ Vaccine is manufactured in compliance with Good Manufacturing Practice (GMP) regulations (21 Code of Federal Regulations [CFR] 21), that is described in detail in Investigational New Drug (IND) 13969. Manufacture of PfSPZ Vaccine is performed in Sanaria s Clinical Manufacturing Facility (CMF) in Rockville, Maryland, USA.
  Arms: Arm 1
Other: PfSPZ Diluent — The diluent for PfSPZ Vaccine is composed of phosphate-buffered saline (PBS) and human serum albumin (HSA) and is termed PfSPZ Diluent (or Diluent). The PfSPZ Diluent was manufactured in compliance with GMP by Sanaria, Inc. (9800 Medical Center Dr., Rockville, MD, USA), or Sanaria s contractor Emergent Biosolutions (https://www.emergentcdmo.com/). Each lot of PfSPZ Diluent is issued a Certificate of Analysis (CoA) and is also placed on a stability program. HSA used in PfSPZ Diluent is a licensed product which is approved for parenteral, IV administration to humans and is purchased by Sanaria, Inc. from CSL Behring, Bern, Switzerland.
  Arms: Arm 1
Drug: Normal Saline — Sterile isotonic (0.9%) normal saline will be procured in the US and shipped to Mali at ambient temperature. Like the study product, normal saline is a clear liquid, making it indistinguishable from the study product when drawn up into a syringe. Normal saline will be used as a placebo, rather than a comparator vaccine being used, as currently there are no licensed vaccines available as IV formulations. The NS to be used in this trial will be an FDA-licensed product which is commercially available (sodium chloride for injection 10 mL by Pfizer). NS will be purchased by Sanaria and supplied to the clinical site.
  Arms: Arm 2

SUMMARY:
Background:

Malaria is a disease that affects many people in Africa. It is caused by germs carried by some mosquitoes. A person bitten by an infected mosquito will get malaria. Most malaria infections cause only mild symptoms or none at all, but sometimes the disease can be deadly. Malaria can also harm pregnant women. They may lose their pregnancies or deliver too early, and the mother and newborn may die. An experimental malaria vaccine (PfSPZ) has shown some protection against malaria infection. It is not yet known if PfSPZ is safe for pregnant women.

Objective:

To test the PfSPZ vaccine in pregnant women.

Eligibility:

Healthy women aged 18 to 34 years at 14 to 32 weeks gestation with 1 fetus.

Design:

The study will be in Mali. Participants will have about 40 clinic visits over 20 months.

They will be screened. They will have an ultrasound exam and a test of their heart function. They will have blood and urine tests.

Participants will receive an injection through a needle into a vein on 3 visits over 1 month. Some will receive the PfSPZ vaccine; others will be injected with salt water. They will not know which injection they are getting.

After the last injection, participants will visit the clinic every 2 weeks. They will have blood tests at each visit.

After giving birth, participants and their infants will visit the clinic every 2 weeks for 4 months; then they will have visits each month until the infant is 1 year old. The infant will be examined and will have blood tests at each visit.

DETAILED DESCRIPTION:
Study Description:

A randomized double blind, placebo-controlled study to assess the safety, tolerability, immunogenicity and protective efficacy of a 1, 8, 29-day regimen of 9x105 PfSPZ of PfSPZ Vaccine or placebo (normal saline) in healthy pregnant women and their fetus/newborn. The first immunization is to be administered at 16 0/7 to 32 6/7 weeks of gestation and targeted to be completed prior to delivery. Offspring and post-partum women will be followed for 12 months post-delivery.

The study is composed of two cohorts (3rd trimester: Arms 1A, 2A, 2nd trimester: Arms 1B, 2B) with two arms (PfSPZ Vaccine, normal saline placebo) and associated offspring. Enrollment and vaccinations will be staggered for safety with only third trimester women (n=30; based on guidance provided by regulatory bodies) enrolling first in two separate subsets (n=10 [5 PfSPZ Vaccine/5 normal saline], n=20 [10 PfSPZ Vaccine/10 normal saline]) and receiving all three doses of vaccine in a staggered manner and undergoing safety reviews prior to further enrollments. Third trimester enrollment in this staggered manner is to account for any significant events occurring immediately post initial vaccinations with the smaller first subset of women (n=10; DSMB review). After all third trimester pregnancy outcomes are reviewed (by DSMB, FDA, Sponsor, EC/IRB), an additional cohort of women in their second trimester will be vaccinated in two separate subsets (n=10 [5 PfSPZ Vaccine/5 normal saline], n=20 [10 PfSPZ Vaccine/10 normal saline]) separated by at least six weeks. A longer time period of review will be conducted during the 2nd trimester out of additional safety measures to ensure no significant events of concern occur post receipt of a full vaccination series (n=10; DSMB review) before proceeding to the last subset of women (n=20).

Arm 1 (9x10^5 PfSPZ Vaccine): (n = 30) pregnant women will receive three doses of PfSPZ Vaccine (9x10^5 PfSPZ) via direct venous inoculation (DVI) at 1, 8, 29 days

* Arm 1A: (n=15) women 28 0/7 to 32 6/7 WGA (third trimester) at time of first vaccination
* Arm 1B: (n=15) women 16 0/7 to 27 6/7 WGA (second trimester) at time of first vaccination

Arm 2 (normal saline): (n = 30) pregnant women will receive normal saline via DVI at 1, 8, 29 days

* Arm 2A: (n=15) women 28 0/7 to 32 6/7 WGA (third trimester) at time of first vaccination
* Arm 2B: (n=15) women 16 0/7 to 27 6/7 WGA (second trimester) at time of first vaccination

All participants will receive intermittent preventive treatment in pregnancy (IPTp) with sulfadoxine-pyrimethamine (SP) as per standard of care in Mali. The study team will coordinate with the women s antenatal care (ANC) provider to time her IPTp prior to vaccine dose 1 (approximately 2 weeks prior) and between vaccine dose 2 and dose 3 (approximately 2 weeks prior to dose 3) within the protocol defined windows.

Pregnant women will be monitored closely for the duration of their pregnancy and for at least 12 months post-partum for safety, tolerability, immunogenicity, and malaria infection during the follow-up period.

Infants (n=up to 60) born to enrolled women will also be monitored closely for 12 months post-delivery for safety, immunogenicity, and malaria infection.

Objectives:

Primary Objectives:

-To describe the safety of PfSPZ Vaccine at 9x10^5 PfSPZ at dosing schedule of 1, 8, 29 days in pregnant women and their fetuses using a composite measure of adverse maternal and birth outcomes

Secondary Objectives:

* To describe the safety and tolerability of PfSPZ Vaccine at 9x10^5 PfSPZ at dosing schedule of 1, 8, 29 days in pregnant women and their fetuses using solicited adverse events (AEs), unsolicited AEs, and laboratory abnormalities
* To describe the safety of maternal vaccination with PfSPZ Vaccine in infants

Exploratory Objectives:

* To explore the protective efficacy against Pf malaria of PfSPZ Vaccine in pregnant women (peripheral blood, placenta) and infants (peripheral, cord blood)
* To assess the immune response to PfSPZ Vaccine in pregnant women and infants and their association with protection against Pf malaria
* To assess genetic relatedness of the PfSPZ Vaccine parasite strain to malaria infection parasites in pregnant women and infants

Endpoints:

Primary Endpoints:

-Composite endpoint of adverse maternal or birth outcomes defined as: preterm birth, miscarriage, stillbirth, early neonatal death, direct maternal death, low birth weight, small for gestational age (counts and proportions)

Secondary Endpoints:

* Safety and tolerability in pregnant women and their fetuses

  * Solicited local and systemic AEs through 7 days post injection (counts and proportions)
  * Clinical laboratory parameters through 14 days post injection (counts and proportions)
  * All unsolicited AEs, AEs of special interest (AESIs), and serious AEs (SAEs) through delivery and six months thereafter (counts and proportions)
* Safety in infants

  * Neonatal SAEs (including late neonatal deaths or AESIs) through 6 months of age (counts and proportions)
  * Growth and developmental milestones through 1 year of age (counts and proportions)
  * All unsolicited AEs through 6 months of age (counts and proportions)

Exploratory Endpoints:

* Protective efficacy

  * Pf blood stage infection measured by blood smear and nucleic acid detection in women starting immediately following 3rd injection over 24-week period (time to event, binary)
  * Pf blood stage infection measured by blood smear and nucleic acid detection in infants through 1 year of age (time to event, binary)
  * Pf blood stage infection measure by blood smear and nucleic acid detection in post-partum women starting immediately following 3rd injection until 1 year post-delivery (time to event, binary)
  * Pf infection measure by blood smear and nucleic acid in cord blood (counts and proportions)
  * Pf infection measure by blood smear and nucleic acid in placentas (counts and proportions)
* Immune responses (antibody, cellular) to PfSPZ Vaccine in pregnant and post-partum women and infants and their association with protection against Pf malaria
* Genotyping of maternal peripheral blood or placental and newborn/infant peripheral or cord blood Pf parasites

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following

criteria:

* Willing and able to provide consent for study participation for herself and for her infant prior to initiation of any study procedures
* Stated willingness to comply with all study procedures and availability of both mother and offspring for the duration of the study
* Healthy, pregnant women 18-34 years of age (inclusive)
* Singleton pregnancy (confirmed by ultrasound)
* Gestational weeks of pregnancy, confirmed by best obstetrical estimate, at minimum of 16 weeks 0 days and a maximum of 32 weeks 6 days of gestation at the time of the first dose of PfSPZ Vaccine and minimum 14 weeks 0 days and maximum of 32 week 0 days of gestation at the time of the first dose of IPTp

  --Note: women may be screened prior to 16 0/7 weeks gestation for dating of pregnancy
* Documented first, second, or third trimester ultrasound with singleton gestation and no significant fetal anomalies or other abnormalities
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
* Identified antenatal care provider outside of the study team
* In good general health as evidenced by medical history
* Willing to have blood samples stored for future research

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this

study:

* Medical, behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol
* Hemoglobin (Hgb), WBC, absolute neutrophils, and platelets outside the local laboratory defined limits of normal per trimester and >= Grade 2 (participants may be included at the investigator s discretion for not clinically significant abnormal values)
* Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined (per trimester) upper limit of normal and >= Grade 2 (participants may be included at the investigator s discretion for not clinically significant abnormal values)
* Infected with HIV, hepatitis B, hepatitis C, syphilis, toxoplasmosis, rubella as documented by testing at screening
* Sickle cell disease (HbSS or HbSC) or sickle trait (HbAS) by testing at screening
* Clinically significant abnormal ECG such as abnormal QTc
* History of receipt of the following:

  * Investigational malaria vaccine in the last 5 years
  * Immunoglobulins and/or blood products within 6 months of enrollment
  * Investigational product within 3 months of enrollment
  * Chronic (>=14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >=20 mg/day or equivalent) or immunosuppressive drugs within 30 days of enrollment
  * Live vaccine within 30 days of enrollment
  * Non-live vaccine within 14 days of enrollment or planned receipt of a killed vaccine within 14 days of scheduled vaccination
* Known medical problems:

  * Pre-existing autoimmune or antibody-mediated diseases (e.g. systemic lupus erythematosus,

rheumatoid arthritis, multiple sclerosis, Sj(SqrRoot)(Delta)gren s syndrome, or autoimmune thrombocytopenia)

* Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past two years, or that has required the use of oral or parenteral corticosteroids at any time during the past two years)
* Immunodeficiency disorder
* Asplenia or functional asplenia
* Diabetes (inclusive of Type 1, 2, or gestational)
* Deep venous thrombosis or thromboembolic event (current or prior history)
* Seizures (exception is simple febrile seizures during childhood)
* History of prior uterine surgery

  * Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies
  * Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
  * History of a severe allergic reaction or anaphylaxis following previous vaccinations or medications
  * Known allergies or other contraindications against: PfSPZ Vaccine, human serum albumin
  * Positive screening testing or diagnostics for entities (pathogens, diseases) deleterious to pregnancy
  * Nullipara (P<1) or grandimultipara (P>=5)
  * Body mass index (BMI) at enrollment >=30
  * Prior or current pregnancy history of:
* 2 or more spontaneous miscarriages
* Any unexplained stillbirths
* Any unexplained neonatal deaths
* Infant with major congenital anomalies
* Infant with known genetic disorder
* Preterm deliveries (< 37 0/7 WGA)
* Severe pre-eclampsia and/or eclampsia
* Gestational hypertension
* Gestational diabetes
* Red blood cell isoimmunization
* Cervical insufficiency or incompetent cervix
* Polyhydramnios or oligohydramnios
* Premature contractions or preterm labor
* Bleeding through gestation
* Known intrauterine fetal growth restriction
* Use of anti-coagulants during pregnancy
* Receipt of progesterone during current pregnancy
* Prior Cesarean section

  * Documentation that current pregnancy results from rape or incest
  * Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the participant unable to comply with the protocol

Max Age: 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety using a composite of adverse maternal and birth outcomes | One year
  Composite endpoint of adverse maternal or birth outcomes defined as: preterm birth, miscarriage, stillbirth, early neonatal death, direct maternal death, low birth weight, small for gestational age (counts and proportions)

SECONDARY OUTCOMES:
Safety and tolerability in pregnant women and their fetuses using solicited adverse events (AEs), unsolicited AEs, and laboratory abnormalities | 7 and 14 days post injection; 6 months after delivery
  Solicited local and systemic AEs through 7 days post injection (counts and proportions) -Clinical laboratory parameters through 14 days post injection (counts and proportions) -All unsolicited AEs, medically attended AEs (MAEs), and serious AEs (SAEs) through delivery and six months thereafter (counts and proportions)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Ou(SqrRoot)(Copyright)less(SqrRoot)(Copyright)bougou, Health Research Center, Ou(SqrRoot)(Copyright)less(SqrRoot)(Copyright)bougou, Mali

IPD SHARING:
Plan to Share IPD: No